CLINICAL TRIAL: NCT02478489
Title: Oral v. Injection Naltrexone in Hospital: Comparative Effectiveness for Alcoholism
Brief Title: Alcohol Disorder hOsPital Treatment Trial
Acronym: ADOPT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-32911; R01AA021335 (NIH)
Record Dates: First submitted 2015-06-11; First posted 2015-06-23 (Estimated); Results first posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Heavy Drinking; Alcohol Dependence; Alcohol Use Disorder
Keywords: alcohol; heavy drinking; naltrexone; hospital; alcohol use disorder; alcohol dependence; comparative effectiveness
MeSH Terms: conditions — Alcoholism | interventions — Naltrexone; vivitrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Extended-release injectable naltrexone (XR-NTX) (Experimental): Monthly XR-NTX (380 mg) Subjects randomized to XR-NTX will receive one intramuscular gluteal injection (in accordance with the FDA approved label/package insert) of 380 mg of NTX for extended-release injectable suspension at study entry (in the hospital) and 1, and 2 months later (outpatient in the primary care clinic), alternating buttocks.
  Interventions: Drug: Extended-release injectable naltrexone (XR-NTX)
- Oral naltrexone (PO-NTX) (Active Comparator): Daily PO-NTX (50 mg, up to 100 mg if heavy drinking continues) Subjects randomized to PO-NTX will receive a study prescription (first one in the hospital)(fillable only at the medical center research pharmacy and prepared by the research pharmacist) for a 1-month supply of oral NTX to be taken once daily- 25 mg a day for 3 days, then 50 mg a day. If the subject has a prior history of taking PO-NTX and tolerating it well, the participant may be started at 50 mg. The dose may be increased to 100 mg daily for any participant who continues to have heavy drinking.
  Interventions: Drug: Oral naltrexone (PO-NTX)

INTERVENTIONS:
Drug: Oral naltrexone (PO-NTX) — oral naltrexone
  Other Names: Revia
  Arms: Oral naltrexone (PO-NTX)
Drug: Extended-release injectable naltrexone (XR-NTX) — injectable naltrexone
  Other Names: Vivitrol
  Arms: Extended-release injectable naltrexone (XR-NTX)

SUMMARY:
The specific aims of this pragmatic randomized controlled trial are to compare initiating injectable extended release naltrexone (XR-NTX) or oral naltrexone (PO-NTX) at the time of discharge from a medical hospitalization for patients with alcohol use disorder (AUD) on: 1) alcohol consumption and consequences, and 2) acute healthcare utilization (including hospital readmission and emergency visits) and cost-effectiveness. In exploratory analyses, the investigators will assess moderators of medication effects including demographic, behavioral, and genetic factors.

DETAILED DESCRIPTION:
Hospitalization for medical illness is a unique and missed opportunity for intervention for alcohol use disorders (AUDs). Referrals can help link patients from hospitals to alcohol treatment. But most patients return to heavy drinking after hospital discharge and do not follow-up with alcohol treatment, risking hospital readmission. Pharmacotherapy has efficacy for AUD, but adherence to these medications is poor. Furthermore, these medications are rarely prescribed in general medical settings, during or after hospitalization. Beginning treatment for AUD during a hospitalization for medical illness could broaden the reach of effective treatment and is likely to be more effective than delaying treatment until a specialist visit or treatment program entry. Hospital discharge is a time of both risk (i.e., for drinking and non-adherence to medical care) and opportunity (i.e., to begin alcohol treatment and complete medical treatments). Interventions that work quickly and improve adherence could improve medical and alcohol-related outcomes.

Oral naltrexone (PO-NTX), and the more-costly-per-dose long-acting injectable extended release naltrexone (XR-NTX) are Food and Drug Administration (FDA)-approved efficacious treatments for AUD. The XR-NTX half-life is 5-10 days and is dosed monthly, whereas the PO-NTX half-life is 13 hours and is dosed daily. The longer half-life of XR-NTX translates into patients receiving effective pharmacotherapy for a longer time without having to adhere to a daily dose. Thus, although more costly per dose, greater effectiveness could mean overall reduced costs of care (including alcohol-related health consequences and healthcare utilization). Despite potential differences in costs and patient preferences, PO-NTX and XR-NTX have not been directly compared in a randomized controlled trial (RCT), they have not been studied as treatments at medical hospital discharge, and their effectiveness in real world practice settings compared with standard care is unknown.

This trial is significant because it will address the clinically relevant comparative effectiveness question and lead to greater adoption of the most effective and cost-effective approach for treating AUD with pharmacotherapy in general hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual of Mental Disorders (DSM) 5 alcohol use disorder (AUD) (assessed using Alcohol Use Disorder and Associated Disabilities Interview Schedule (AUDADIS))
* ≥1 heavy drinking episodes (≥5 standard drinks [4 for women] in a day) in 30 days prior to hospitalization*
* Inpatient on a hospital general medical service
* Adult (age 18 years or greater)
* Ability to speak English (fluency)
* ≥2 contact persons*

Exclusion Criteria:

* Pregnancy (urine testing if childbearing potential)
* Currently breast-feeding
* Urine expanded panel drug test (dipstick) positive for opiates, semi-synthetic or synthetic opioids
* Opioid use (self-report and verification in medical record) in past 7 days for long-acting opioids
* Opioid use in past 24 hours for short-acting opioids
* Discharge prescription for opioids
* Future need for opioids for an anticipated painful event or surgery
* Known hypersensitivity to NTX
* Acute severe psychiatric illness (currently suicidal or psychotic)
* Cognitive dysfunction that precludes informed consent or research assistant (RA) assessment that subject cannot understand interview questions
* Alanine aminotransferase or aspartate aminotransferase >5 times the upper limit of normal
* Acute hepatitis
* Liver failure
* Known severe thrombocytopenia (<50,000)
* Coagulopathy
* Coagulation disorder
* Body habitus that precludes intramuscular injection
* Plans to leave the Boston area in less than one year
* Enrollment in a research study which involves taking a pharmaceutical agent that is expected to interact with naltrexone

[*criteria not changed since study start; change reflects correction of typo]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Saitz, MD, MPH, Principal Investigator — Boston University
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The ADOPT study dataset will include data from 260 subjects, including self-reported demographic and alcohol/drug use information as well as study-specific assessments and information obtained from urine and blood samples. All IPD and sample repository data will be made available to interested and qualified researchers wishing to conduct secondary analyses of the data. The final datasets will be stripped of identifiers prior to release for sharing.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: IPD will first be available to ADOPT study investigators and Boston Medical Center and Boston University affiliated trainees. After establishing the specific areas to be addressed in the papers reporting the main findings of the study, all IPD and sample repository data will be made available for sharing starting 12 months after publication of these main study findings.
Access Criteria: The ADOPT study PI (Saitz), with co-investigator consultation as necessary, will review and approve proposals submitted by interested and qualified researchers wishing to conduct secondary analysis of the data and use of biological samples beyond the main planned reports of study findings. If proposals are approved, the investigators will make the de-identified IPD and samples available for analysis, provided IRB approval is obtained. These investigators will be provided with study forms and documents (e.g., data dictionary, procedure manuals, study questionnaires as appropriate) that allow accurate understanding of the datasets. Costs associated with data sharing will be the responsibility of investigators seeking the data.

REFERENCES:
- [Derived] Magane KM, Dukes KA, Fielman S, Palfai TP, Regan D, Cheng DM, Lee H, Kraemer KL, Bullard MJ, Chen CA, Samet JH. Oral vs Extended-Release Injectable Naltrexone for Hospitalized Patients With Alcohol Use Disorder: A Randomized Clinical Trial. JAMA Intern Med. 2025 Jun 1;185(6):635-645. doi: 10.1001/jamainternmed.2025.0522. PMID 40257810

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Extended-release Injectable Naltrexone (XR-NTX) | Oral Naltrexone (PO-NTX)
Started | 123 | 125
Completed | 108 | 109
Not Completed | 15 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Extended-release Injectable Naltrexone (XR-NTX) | Oral Naltrexone (PO-NTX) | Total
Number analyzed (Participants) | 123 | 125 | 248
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.4 (10.3) | 49.4 (10.5) | 49.4 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 25 | 49
  Male | 99 | 100 | 199
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 19 | 39
  Not Hispanic or Latino | 103 | 106 | 209
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 10 | 3 | 13
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 3 | 2 | 5
  Black or African American | 61 | 64 | 125
  White | 47 | 54 | 101
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Percent heavy drinking days over the past 30 days assessed at baseline by Timeline Followback [Mean (Standard Deviation); unit: Percent heavy drinking days of past 30] | 70.7 (31.5) | 66.7 (31.5) | 68.7 (31.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Percent Heavy Drinking Days (%HDDs) Over the Past 30 Days From Baseline to 3 Month Follow-up, Assessed Using the Timeline Follow-Back
Description: The primary alcohol use outcome will be change in percent heavy drinking days (%HDDs) from baseline to 3 month follow-up. %HDDs out of the past 30 days is assessed using the Timeline Follow-Back. %HDDs is the most likely (and most sensitive) to be affected by NTX and is clinically important (any reduction means less risk of harm). We chose self-report because biological testing is not sufficiently valid for detecting drinking levels and changes of clinical importance. The self-report tool is valid, particularly so when staff are well trained, and when the context for the subject is: they are informed they are being tested for consumption (breath alcohol and carbohydrate deficient transferrin (CDT), there are no consequences related to consumption levels, and that results are being recorded confidentially.
Time Frame: Baseline, 3 months
Population: Analysis population includes those who completed the 3 month follow-up assessment. Population does not match baseline sample due to attrition / loss to follow-up.
Measure: Mean (Standard Deviation); unit: change in percent heavy drinking days
Arm/Group | Extended-release Injectable Naltrexone (XR-NTX) | Oral Naltrexone (PO-NTX)
Number analyzed (Participants) | 108 | 109
change in percent heavy drinking days | -46.4 (38.5) | -38.4 (43.3)

2. Secondary Outcome: Acute Care Hospital Utilization
Description: Any acute hospital utilization (emergency department visit or inpatient stay) over the past 90 days assessed at 3-month follow-up by the Form 90. Self-report for short-term high impact, memorable health utilization such as emergency and hospital stays is valid and can measure utilization at any site. Using the clinical data warehouse at one site (Boston Medical Center (BMC)) and statewide data, we will compare self-report to the utilization databases. But, self-report data will remain primary, with databases used to provide a descriptive frame of reference.
Time Frame: 3 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Extended-release Injectable Naltrexone (XR-NTX) | Oral Naltrexone (PO-NTX)
Number analyzed (Participants) | 108 | 109
Participants
  Any acute care hospital utilization (emergency department visit or inpatient stay) | 66 | 59
  No acute care hospital utilization (emergency department visit or inpatient stay) | 42 | 50

3. Other Pre Specified Outcome: Medication Adherence
Description: High adherence to XR-NTX will be defined as administration of XR-NTX by the study nurse 3 times. Medium adherence will be defined as 1 or 2 injections. For PO-NTX, high adherence will be defined as participant self-report of taking PO-NTX for 90 out of the past 90 days at the 3 month study visit, and medium adherence as participant self-report of taking PO-NTX for 30-89 out of the past 90 days at the 3 month study visit (Form 90). We will also assess the presence of detectable beta-naltrexol to confirm reports of recent pill taking.
Time Frame: 1, 2 and 3 months
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Alcohol Consequences Via Questionnaire
Description: Alcohol consequences over the past 3 months will be measured by collecting participant self-report data via the Short Inventory of Problems (SIP-2R) at 3-month follow-up. The SIP-2R is a validated 15-item measure for assessing recent adverse consequences associated with alcohol use.
Time Frame: 3 months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Alcohol Use Disorder-related Treatment Utilization Via Questionnaire and Health Records
Description: Alcohol use disorder-related treatment utilization over the past 90 days assessed at 3-month follow-up by the Form 90. Using the clinical data warehouse at one site (Boston Medical Center (BMC)) and statewide data, we will compare self-report to the utilization databases. But, self-report data will remain primary, with databases used to provide a descriptive frame of reference.
Time Frame: 3 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Cost Via Utilization Questionnaire, Health Records and Estimates From Local and National Sources
Description: Healthcare utilization cost data will be collected via the Form 90 for self-reported outpatient and emergency visits, hospitalizations, and specialty addiction treatment. Utilization episodes will be converted to costs by use of Medicare relative value units (RVUs) for acute inpatient care, Resource Based Relative Value System (RBRVS) units for Medicare reimbursement of outpatient visits, and the average daily rate for long-term care.
Time Frame: 3 and 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Events were collected until the participant's 3-month follow-up research assessment was completed or their follow-up window closed.
Arm/Group | Extended-release Injectable Naltrexone (XR-NTX) | Oral Naltrexone (PO-NTX)
All-Cause Mortality (participants affected / at risk) | 2/123 | 3/125
Serious Adverse Events (participants affected / at risk) | 43/123 | 43/125
Other Adverse Events (participants affected / at risk) | 59/123 | 39/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Extended-release Injectable Naltrexone (XR-NTX) (N=123) | Oral Naltrexone (PO-NTX) (N=125)
Abdominal Pain (Gastrointestinal disorders) | 1 | 4
Acute Cholecystitis (Hepatobiliary disorders) | 0 | 1
Alcohol Withdrawal (Psychiatric disorders) | 6 | 10
Altered Mental Status (Nervous system disorders) | 1 | 0
Ankle Fracture (Musculoskeletal and connective tissue disorders) | 0 | 2
Ankle Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal Ganglia Hemorrage (Nervous system disorders) | 1 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cellulitis (Skin and subcutaneous tissue disorders) | 0 | 1
Chest Pain (Cardiac disorders) | 1 | 4
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Congestive Heart Failure (Cardiac disorders) | 2 | 1
Coronavirus (COVID-19) (Infections and infestations) | 0 | 1
Death (General disorders) | 2 | 3
Depression (Psychiatric disorders) | 0 | 1
Diabetic Ketoacidosis (Endocrine disorders) | 1 | 2
Dizziness (Nervous system disorders) | 1 | 0
Epigastric Pain (Gastrointestinal disorders) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 2 | 1
Fatigue (General disorders) | 1 | 0
Foot Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Hallucinations (Psychiatric disorders) | 0 | 1
Heart Failure (Cardiac disorders) | 1 | 0
Hyperglycemia (Endocrine disorders) | 0 | 2
Hypertension (Cardiac disorders) | 1 | 0
Hypoglycemia (Endocrine disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hypotension (Cardiac disorders) | 1 | 0
Injection Site Abscess (Skin and subcutaneous tissue disorders) | 1 | 0/0
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Intoxication (Injury, poisoning and procedural complications) | 3 | 0
Laparoscopic Cholecystectomy (Surgical and medical procedures) | 0 | 1
Left Hand Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Lower Extremity Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteomylelitis of Toe (Infections and infestations) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 2
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Psychiatric Hospitalization (Psychiatric disorders) | 1 | 0
Pulmonary embolism (Vascular disorders) | 1 | 0
Rectal Bleeding (Gastrointestinal disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Seeking Detox (Psychiatric disorders) | 1 | 0
Seizure (Nervous system disorders) | 5 | 2
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Subdural Hematoma (Nervous system disorders) | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 1 | 2
Suicide Attempt (Psychiatric disorders) | 1 | 1
Syncope (Cardiac disorders) | 3 | 1
Thoracic Osteomyelitis (Nervous system disorders) | 0 | 1
Traumatic Injury (Injury, poisoning and procedural complications) | 1 | 0
Urinary Tract Infection (Renal and urinary disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 3
Weakness (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Extended-release Injectable Naltrexone (XR-NTX) (N=123) | Oral Naltrexone (PO-NTX) (N=125)
Elevated Liver Function Tests (Hepatobiliary disorders) | 19 | 32
Injection Site Discomfort (Skin and subcutaneous tissue disorders) | 36 | 0/0
Intoxication (Injury, poisoning and procedural complications) | 16 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-24): https://cdn.clinicaltrials.gov/large-docs/89/NCT02478489/Prot_SAP_000.pdf